CLINICAL TRIAL: NCT01325363
Title: Novel Metaphor Processing Among Schizophrenic Patients - Magnetoencephalographic (MEG) Evidence
Brief Title: Magnetoencephalographic (MEG) Evidence for Novel Metaphor Processing Among Schizophrenic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHA-11-0006
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Novel Metaphor
Keywords: Schizophrenia; Novel metaphor
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schizophrenia (Experimental): Schizophrenic patients
  Interventions: Device: Magnetoencephalograph (MEG)
- Control (Experimental): Neurotypical subjects
  Interventions: Device: Magnetoencephalograph (MEG)

INTERVENTIONS:
Device: Magnetoencephalograph (MEG) — Brain imaging device that records the magnetic fields in the brain.
  Other Names: MAGNES STIMULUS, 4-D NEUROIMAGING, 9727 Pacific heights blvd., San Diego, CA 92121, USA.

SUMMARY:
The aim of this research is to investigate the neurolinguistic mechanisms underlying thought disorders among schizophrenic patients. In particular, it will investigate the neurolinguistic basis for loose association - a phenomena which this population is characterized by. Several researchers have previously suggested that loose associations among schizophrenic patients relate to a lack of inhibition in the automatic spread of activation mechanisms within semantic networks (e.g., Soriano, Jimenez, Roman, & Bajo, 2008). This research focuses on the relationship between I. the left-right hemisphere dynamic and II. semantic processing, among schizophrenic patients. The research follows Jung-Beeman's (2005) model which relates semantic associations, activation and inhibition processes to the functioning of the two cerebral hemispheres.

Previous research suggests that, when compared to the neurotypical population, people with schizophrenia show a less defined - or even reversed - hemispheric lateralization pattern for semantic processing. This is linked to an impairment in language function in the left hemisphere, and to a language functions shift from left to right hemisphere (e.g., Crow, 1997). The investigators assume that this unique lateralization pattern may cause a change in balance in the semantic activation and inhibition system among schizophrenic patients.

As stated, one of the linguistic models that predicts how reduced left hemisphere dominancy will influence linguistic functioning is Jung-Beeman's (2005) bilateral model for language understanding. According to this model, the left hemisphere specializes in precise and fine semantic processing, while the right hemisphere specializes in coarse and abstract semantic processing. Building upon this distinction, our assumption is that schizophrenic patients experience a difficulty in fine semantic processing which is caused by functional impairment in the left hemisphere. It is our further assumption that coarse semantic processing - located in the right hemisphere - is relatively unimpaired. This change in the balance between the two processes may have direct implications on the associative semantic network among schizophrenic patients.

In order to test this hypothesis, the current research will make use of a specific language expression type which involves fine and coarse semantic processing, and for which there is evidence for crucial right hemisphere involvement: novel metaphor processing. 10-20 adult schizophrenic patients will be presented with four different types of two word expressions: literal; conventional metaphor; novel metaphor and unrelated. The patients will have to decide as quickly and accurately as possible if the expression is meaningful or meaningless while their brain activity is recorded by a Magnetoencephalographic (MEG) device (which combines a high temporal resolution with the ability to localize the activity).

Therefore, our main hypothesis is that schizophrenic patients will show a bilateral brain activity pattern when conducting semantic decisions, and that this pattern will be related to improved reaction times and accuracy when presented with novel metaphors than when presented with other types of expressions.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic patients according to Diagnostic and Statistical Manual of Mental Disorders (DSM IV) or International Classification of Diseases (ICD-10)
* Hebrew native speakers

Exclusion Criteria:

* Language disabilities
* Left handed
* Reading disabilities
* Brain damage
* Impaired intelligence
* Metal implants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Amplitude power and source location of the magnetic brain activity | one hour
  Magnetic brain activity which was recorded during the experimental task, will be cleaned from artifacts, averaged over participants and then the amplitude power of each condition in each group will be calculated for different time windows. In a subsequent analysis, the source location of the activity will be calculated using Beamforming techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- shalvata MHC, Hod HaSharon, Israel